CLINICAL TRIAL: NCT01073917
Title: Effects of Spontaneous Breathing Activity on Atelectasis Formation During General Anaesthesia: A Randomized Clinical Trial
Brief Title: Effects of Spontaneous Breathing Activity on Atelectasis Formation During General Anaesthesia
Acronym: SBAFGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Oliver C. Radke, MD, PhD, DEAA, Dpt. of Anesthesia and Intensive Care Medicine, University Hospital, TU Dresden, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EK375122009
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Atelectasis
Keywords: Ventilation; General Anesthesia; electrical impedance tomography; pressure support; spontaneous breathing; laryngeal mask; Patients who are scheduled for elective knee or ankle surgery
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Spontaneous Breathing (Other): Patients will be breathing spontaneously during anesthesia
  Interventions: Other: Spontaneous Breathing
- Pressure controlled ventilation (Other): Patients in the PPV group will be ventilated by pressure control (tidal volume 8-10 ml/kg, frequency 10-14, I:E 1:1, no PEEP, target CO2 4.5 kPa).
  Interventions: Other: Pressure Controlled Ventilation
- Pressure Support Ventilation (Other): The patients in the PSV group will breathing spontaneously on the ventilator with assistance by inspiratory support pressure. The support pressure will be adjusted to achieve a tidal volume of 8-10 ml/kg.
  Interventions: Other: Pressure Support Ventilation

INTERVENTIONS:
Other: Spontaneous Breathing
  Arms: Spontaneous Breathing
Other: Pressure Controlled Ventilation
  Arms: Pressure controlled ventilation
Other: Pressure Support Ventilation
  Arms: Pressure Support Ventilation

SUMMARY:
Atelectasis and redistribution of ventilation towards non-dependent lung zones are a common side effects of general anesthesia. Spontaneous breathing activity (SBA) during mechanical ventilation may avoid or reduce atelectasis, improving arterial oxygenation; however, it is unclear whether these effects play a significant role during general anesthesia in patients with healthy lungs. Earlier studies on ventilation during general anesthesia had to rely on computed tomography (CT) findings. Recent advances in lung imaging technology allow to assess the regional aeration of the lungs continuously and non-invasive by electrical impedance technology (EIT). In this work, we will use the EIT to assess ventilation changes from the time before induction of anesthesia until discharge from the post-anesthesia care unit. Our main focus is the difference caused by pure positive pressure ventilation (PCV) and assisted spontaneous breathing (pressure support ventilation, PSV). Our findings would improve our understanding of the physiology of the lungs during general anesthesia and would help to improve the standards of respiratory care during anesthesia

DETAILED DESCRIPTION:
Atelectasis formation is a common phenomenon during general anaesthesia, occurring in almost 90% of patients (Lundquist, Hedenstierna et al. 1995). In patients in supine position, atelectasis of dorsal lung zones is usually accompanied by redistribution of ventilation towards ventral areas (Hedenstierna 2003; Victorino, Borges et al. 2004).The main mechanisms which contribute to the formation of atelectasis are compression (e.g. in obese patients or during laparoscopic surgery), absorption (e.g. when high concentrations of inspired oxygen are used) and reduced surfactant action(Magnusson and Spahn 2003). Atelectasis impairs oxygenation by reducing the functional residual capacity and by causing right-to-left-shunts. Consecutively, hypoxemia after extubation is common in daily practice: 20% of patients in a study experienced desaturations below 92% (Mathes, Conaway et al. 2001), and the risk is even higher in patients with risk-factors such as obesity or thoraco-abdominal procedures (Russell and Graybeal 1993; Xue, Li et al. 1999). Hypoxemic events prolong the stay in PACU, cause more ICU admissions and increase the incidence of cardiac complications (Rosenberg, Rasmussen et al. 1990; Gill, Wright et al. 1992).

Several measures to prevent or treat atelectasis in ventilated patients have been investigated, such as PEEP (Brismar, Hedenstierna et al. 1985; Tokics, Hedenstierna et al. 1987; Neumann, Rothen et al. 1999), recruitment maneuvers (Neumann, Rothen et al. 1999) and spontaneous breathing during mechanical ventilation (Putensen, Rasanen et al. 1994; Putensen, Mutz et al. 1999). The laryngeal mask airway (LMA) is ideally suited for spontaneous breathing during general anaesthesia because of its low resistance. A large survey found that more than half of the routine cases with an LMA are performed under spontaneous ventilation (Verghese and Brimacombe 1996), while positive pressure ventilation is equally acceptable. With regard to the prevention of atelectasis, spontaneous ventilation could be advantageous.

Most works on atelectasis formation during general anaesthesia used CT. Although CT is a gold standard for quantification of lung aeration, it can only provide data on single time points and is not suitable for measurements during routine cases. In recent years, the electrical impedance tomography (EIT) has evolved into a versatile tool, which allows detailed insights into ventilation and perfusion conditions of the lung (Bodenstein, David et al. 2009). EIT allows continuous assessment of lung aeration, is non-invasive and can easily be used as a research and monitoring tool during routine cases.

We hypothesize that compared with positive pressure ventilation (PPV), pressure support ventilation (PSV) during general anaesthesia reduces the extent of redistribution as detected by EIT during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 18-65) scheduled for elective knee or ankle surgery under general anaesthesia with an LMA with an expected duration of at least 60 minutes.

Exclusion Criteria:

* Pregnancy,
* Pulmonary diseases (e.g. Asthma, COPD),
* Implanted pacemaker or AICD,
* Inability to communicate or understand the risks of the study,
* Contraindications for an LMA (e.g. obesity, reflux),
* Deformities of the thorax,
* Failure to place an LMA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Regional ventilation at the end of anaesthesia and at discharge from PACU compared to baseline values obtained before induction | Before, during and after anesthesia

SECONDARY OUTCOMES:
Differences in spirometry values, oxygenation in the PACU (measured as SpO2 at room air), breathing effort | Before, during and after anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Carl-Gustav-Carus, Dresden, Saxony, Germany

REFERENCES:
- See also: Department of Anesthesia and Intensive Care Medicine, University Hospital Dresden, Germany — http://anaesthesie-dresden.de/